CLINICAL TRIAL: NCT07107100
Title: Comparison of Periodontal Health, Bonding Time and Failure Between Direct and Indirect Fixed Retainer Placement Among Orthodontic Patients - A Modified Split-mouth Randomized Controlled Trial
Brief Title: Comparison of Periodontal Health, Bonding Time and Failure Between Direct and Indirect Fixed Retainer Placement Among Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Rashna Hoshang Sukhia, Associate Professor, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-9292-32612; 375 (Other Grant/Funding Number: MBBS '88 Student and Trainee Initiated Research)
Record Dates: First submitted 2025-07-12; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Orthodontic Treatment
Keywords: fixed retainer, retainer breakage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Other): those in which fixed retainer is placed using conventional method
  Interventions: Other: a silicon jig/key is used to place/bond fixed retainer on teeth
- Silicon Jig (Experimental): those in which fixed retainer was placed using a silicon jig
  Interventions: Other: a silicon jig/key is used to place/bond fixed retainer on teeth

INTERVENTIONS:
Other: a silicon jig/key is used to place/bond fixed retainer on teeth — a silicon jig/key is used to place/bond fixed retainer on teeth

SUMMARY:
The placement technique of retainers in both maxillary and mandibular arches can influence the time taken for bonding the retainer in the mouth of a patient which can in turn affect the patient´s response to the procedure. The different placement techniques can influence the stability of the retainer wire on teeth and the maintenance of periodontal health during the retention period. Therefore, it is essential to know which technique is better suited for placement and its influence on periodontal health so that in the future it helps clinicians save their time during placement of retainers while benefiting the patients. To our knowledge, this will be the first study both locally and internationally that will include an assessment of periodontal health, time duration of placement and stability of fixed retainer in the maxillary arch as well. Three months period is sufficient for assessment of periodontal health and failure of retainer, long term studies can be at a risk of attrition bias.

OBJECTIVES:

The objectives of this study are:

* The primary objective of this study is to compare the failure of fixed retainers, along with periodontal health and bonding time, which are bonded either through direct method or indirect method on patients undergoing orthodontic debonding through a modified split-mouth technique using mean values for plaque index, gingival index, calculus index follow up appointments over a period of three months.
* The secondary objective of the study is to assess the amount of time taken during placement of retainers via both direct and indirect bonding of fixed retainers

DETAILED DESCRIPTION:
HYPOTHESIS:

* Null Hypothesis: There is no difference in placement technique of fixed retainers that can influence the failure of fixed retainers.
* Alternate Hypothesis: There is a 54% difference in placement technique of fixed retainers that can influence the failure of fixed retainers.

MATERIAL & METHODS:

Study Design: A modified split-mouth randomized controlled trial Settings: Department of Surgery, Dental clinics at the Aga Khan University Hospital.

Study Duration: Minimum six months after ethical review committee (ERC) approval, two months will be used for recruitment of participants in this study.

SAMPLE SIZE:

The size of sample was measured using Open-epi software by using the findings of Gokce et al.15, keeping α as 5%, the power of study as 80% and confidence level at 95%. To calculate sample size, the investigators used the mean and standard deviation values of gingival index at one week interval (0.54 ± 0.64) and (1.02 ± 0.67) for two different bonding techniques i.e direct and indirect, of fixed retainer placement. A sample size of 30 was achieved in each group accounting for the total sample size of 60.

Sampling Technique: Non-probability consecutive sampling

Sample Selection:

Inclusion Criteria:

* Patients aged between 18 - 40 years
* Patients who read, write and understand English language
* Patients undergoing fixed orthodontic treatment
* Patients with good oral hygiene, with grade 1 or below on plaque and gingival indices at the time of debonding of brackets.
* All patients who will sign the informed consent form

Exclusion Criteria:

* Patients with periodontal disease
* Patients with any systemic disease
* Pregnant or nursing females
* Patients who cannot come for follow up appointments for a retainer check up

DATA COLLECTION PROCEDURE:

Before the initiation of the study, ethical approval will be taken from the institutional Ethical Review Committee of AKUH. This study will be carried out as per guidelines of the World Medical Association's Declaration of Helsinki and the principles of Good Clinical Practice (GCP). Any modifications in the protocol will be re-submitted to the ERC. The study will be conducted in compliance with regulations and a copy of the final study protocol will be submitted to ERC. All participants will be given the choice to either accept or refuse their inclusion in the study after providing them with complete detailed information. Only those patients signing the informed consent (Annexure E) will be recruited as study participants. All the data recorded of patients will remain confidential. Access will be provided to no one except the investigators. Participants' names and identities will remain undisclosed; however, data may be seen by ERC or any local regulatory body. Data will be saved for 15 years as per regulatory requirements and institutional guidelines.

Participants will be assigned to one of the two study groups using a computer-generated randomization list using a random permuted block sampling of 6. The investigators of the study will not be blinded. The recruitment of the patients will be performed by the investigator who will explain the objective, the two arms of the study and the allocation to the participants. Patients will be recruited by principal investigator Dr. Rashna and co-investigator Dr. Fizzah on the basis of the above-mentioned inclusion and exclusion criteria. A proper thorough history and examination will be taken by the principal investigator and co-investigator for the purpose of appropriate recruitment of patients. Sequentially numbered, opaque, sealed envelopes method will be implemented for allocation concealment, which will conceal the sequence until interventions are being assigned. Allocation of one of two retainer placement techniques will be assigned using closed sealed envelopes. Randomization will be done by closed sealed envelopes. The randomization will be performed by CTU. The study investigators and patients will not be blinded. The eligible upper and lower arches in each subject will be randomized to one of two groups at a 1:1 allocation ratio. Randomization will aid in minimizing selection bias. Envelopes must be stored in a secure place and opened one by one, only after the subject has been found eligible to be randomized.

A fixed retainer wire will be placed either through direct method or indirect method on randomely selected either of the maxillary and mandibular teeth of orthodontic patients after debonding procedure. All the measurements will be recorded by the investigator on a plaque index (Annexure A), gingival index (Annexure B) and calculus index (Annexure C).

Data will be collected on an organized study proforma (Annexures D). The patients will be recruited from the Dental clinics, AKUH. All patients who will sign the informed consent form (Annexure E) will receive detailed information regarding the study. Data will be collected at three points in time. First, at the time of placement of retainer (T-0), their periodontal health will be recorded on the chart using the plaque, calculus and gingival indices and bonding time will be recorded using a timer. At the follow-up appointments at 1 month (T-1), 3 months (T-2), retainer breakage, gingival and periodontal health findings will be assessed clinically.

Study groups:

The patients will be screened using the inclusion and exclusion criteria by the investigator. Plaque will be assessed using a Community Index of Periodontal Treatment Needs (CPITN) probe before bonding at T-0, T-1, and T-2. Measurements will be taken for the plaque and gingival indices and bonding time will be assessed using a timer. Retainer failures and periodontal health will be assessed at the follow-up appointments.

Group A (Intervention): Indirect placement of retainer (first making of retainer in lab and then it´s transfer from the cast onto the teeth via silicon key.) Group B (Control): Direct placement of retainer ( no prior lab work). The participants will receive routine instructions for oral hygiene maintenance and care of the appliance verbally.

The investigator will unseal the envelope from the CTU, containing information regarding the intervention to be used on the participants based on randomization.

Retainers' management:

Routine oral hygiene maintenance and retainer management instructions will be given to each recruit. The participants will be advised to not bite from their front teeth as it may make retainer wire susceptible to breakage. In case, patient feels wire has moved, tooth has moved or wire is hindering chewing and irritating soft tissues such as tongue, gingiva, patients are advised to report to orthodontic clinics for timely repair of retainer wire.

Interim Analysis/ Stopping Rules:

Interim analysis will be run once after achievement of data collection of 50% of sample size. On the basis of results, it will be decided whether the study will be continued. In case of more than 54% significant difference in failure of fixed retainers, and significant difference in periodontal health and bonding time in two different bonding techniques of fixed retainers, the study will be stopped.

DATA ANALYSIS:

Data will be entered and analyzed in SPSS for Windows (version 23.0, SPSS Inc. Chicago). Frequencies and proportions will be reported for categorical variables such as gender. The Shapiro-Wilk test will be used to check the normality of the data. Descriptive statistics, such as means and standard deviations for normally distributed or median and interquartile range (IQR) for non-normally distributed data will be reported for all baseline clinical factors such as age, gender, type of malocclusion, duration of retainer placement since two different methods are used. Further, gingival and periodontal health may modify/effect the survival of retainers. Repeated measures Anova will be used for the pairwise comparison at baseline, one month and two months follow up. Independent sample t-test will be used for the comparison between the two groups to compare the values between both groups at T-0, T-1, and T-2. Univariate Cox regression analysis will be used to assess the influence of factors such as age, gender, and type of malocclusion on periodontal health and retainer failures. Significant variables at univariate level will be taken to the multivariable regression. Cox proportional hazard regression will be run for survival analysis to assess the survival time of both, DB and IDB. The significance level will be kept at p ≤ 0.05 and confidence level will be kept at 95%.

Data management and confidentiality:

Confidentiality regarding patient information will be strictly followed. Except investigators nobody will have access to patient information. There will be no disclosure at any time of participants' name and identity. However, the data may be seen by ERC, or any local regulatory body for monitoring and audit purpose. As per GCP and other guidelines, data will be retained for 10 years.

Publication policy/plan:

For publication, the anonymized data will be utilized, and it could be presented in either national or worldwide forum.

Data monitoring and quality assurance:

Study PI will randomly check the data for accuracy and completeness on ongoing basis.

Ethical considerations:

Before the initiation of the study, ethical approval will be taken from the institutional Ethical Review Committee of AKUH. This study will be carried out as per guidelines of the World Medical Association's Declaration of Helsinki and the principles of Good Clinical Practice (GCP). Any modifications in the protocol will be re-submitted to the ERC. The study will be conducted in compliance with regulations and a copy of the final study protocol will be submitted to ERC. All participants will be given the choice to either accept or refuse their inclusion in the study after providing them with complete detailed information. Only those patients signing the informed consent (Annexure E) will be recruited as study participants. All the data recorded of patients will remain confidential. Access will be provided to no one except the investigators. Participants' names and identities will remain undisclosed; however, data may be seen by ERC or any local regulatory body. Data will be saved for 10 years as per GCP and institutional guidelines.

Possible risks or benefits:

There is a risk of breakage of retainer wire. In case of retainer breakage, there can be a risk of flexible retainer wire irritating the gums and hinder chewing and for this reason patients are advised to come to dental clinics for timely repair of retainer wire.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 - 40 years
* Patients who read, write and understand English language
* Patients undergoing fixed orthodontic treatment
* Patients with good oral hygiene, with grade 1 or below on plaque and gingival indices at the time of debonding of brackets.
* All patients who will sign the informed consent form

Exclusion Criteria:

* Patients with periodontal disease
* Patients with any systemic disease
* Pregnant or nursing females
* Patients who cannot come for follow up appointments for a retainer check up

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Assessment of retainer failure | 3 months with 3 follow ups, one at the time of placement and one at 1 month, next on 3rd month
  using the frequency of breakage of retainer wire, we will assess retainer failure

CONTACTS AND LOCATIONS:
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
In order to assess outcomes, only the retainer breakage frequency, gingival health scores on an organised proforma will be shared between principal and sub investigators
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: august 2025 till december 2025
Access Criteria: Principal Investigator

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT07107100/Prot_SAP_ICF_000.pdf